CLINICAL TRIAL: NCT00991562
Title: An Open-Label Phase I Study of Bb-10901 (IMGN901, huN901-DM10 in Combination With Lenalidomide and Dexamethasone in Patients With CD56-positive Relapsed or Relapsed/Refractory Multiple Myeloma
Brief Title: IMGN901 in Combination With Lenalidomide and Dexamethasone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMGN0005
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Myeloma
Keywords: relapsed or relapsed/refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — lorvotuzumab mertansine; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: IMGN901 — dose escalation study. dosing on days 1, 8 and 15 every 28 days
  Other Names: BB-10901; huN901-DM1

SUMMARY:
The purpose of this study is to test IMGN901 in combination with lenalidomide and dexamethasone every 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma based on standard criteria.
* Patients must have CD56-positive, relapsed or relapsed/refractory multiple myeloma. Myeloma is considered CD56-positive if either immunohistochemistry (IHC) or flow cytometry criteria defined in Appendix X are met.
* Age < 18 years at the time of signing Informed Consent.
* Patients have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* During the dose escalation phase, patients must have received at least one prior therapy for multiple myeloma. The prior therapy or therapies can include lenalidomide treatment.
* Once the MTD/RPTD is defined, only patients who have received at least 1 but no more than 3 prior chemotherapy regimens will be enrolled at this dose level in the study. Prior regimen(s) may have included bortezomib or a bortezomib component. If prior regimen(s) included a lenalidomide component:

  * Patients last dose of lenalidomide must be ≥ 6 months from Day 1 treatment with BB-10901 (with the exception of maintenance lenalidomide treatment which should be completed at least 4 weeks prior to Day 1 treatment with BB-10901) ,
  * Patients must have achieved a response of stable disease or better to any lenalidomide treatment, and
  * Patients must not have discontinued treatment due to lenalidomide intolerance.
* Patients must be able to adhere to the study visit schedule and other protocol requirements.
* Patients must understand and voluntarily sign an informed consent document.
* Woman of child bearing potential (WCBP) must have a negative pregnancy test within 10 - 14 days and within 24 hours prior to writing an initial prescription for lenalidomide even if continuous abstinence is the chosen method of birth control. In addition, all sexually active WCBP must agree to frequent pregnancy tests as outlined in the protocol and must agree to use 2 contraceptive methods. WCBP must agree to follow these requirements for at least 4 weeks before beginning treatment with lenalidomide and for at least 4 weeks after the last treatment of lenalidomide.
* Male patients must agree to use a latex condom even if he has had a successful vasectomy and males can not donate sperm. Males must agree to follow these requirements for at least 4 weeks following last dose of study drug.
* Patients may have received chemotherapy or wide-field radiotherapy (e.g. .30% of marrow-bearing bones) if completed at least 4 weeks prior to Day 1, or focal radiation completed at least 2 weeks prior to Day 1, and the patient has recovered or stabilized from all adverse effects of such therapy. Therapy with nitrosoureas or mitomycin C must be completed 6 weeks prior to Day 1. Major surgery (this does not include placement of vascular access device or tumor biopsies) must be completed 4 weeks prior to Day 1. Antineoplastic therapy with biological agents must be completed at least 2 weeks prior to Day 1.
* Absolute neutrophil count (ANC) ≥ 1000 cells/mm3, hemoglobin ≥ 8.5 g/dL, and platelet count ≥ 50,000/mm3
* Aspartate aminotransferase(AST) (serum glutamic oxalacetic transaminase, SGOT) and alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase, SGPT) ≤ 3 x upper limit of normal (ULN) and total bilirubin ≤ 1.5 x ULN
* Amylase and lipase levels must be ≤ 1.5 x ULN.
* Serum Creatinine ≤ 1.5 x ULN
* Left ventricular ejection fraction ≥ lower limit of normal (LLN) on MUGA scan or ECHO.
* Patients must agree to follow all guidelines from the RevAssist® Program

Exclusion Criteria:

* Concomitant therapy with other antineoplastic treatments (chemotherapy, radiotherapy or biological agents) during the study.
* Peripheral neuropathy of grade 2 or greater.
* Known hypersensitivity to lenalidomide or other thalidomide derivatives, previous monoclonal antibody therapy or maytansinoids.
* History of deep venous thrombus or pulmonary embolism within 6 months of study enrollment.
* Any serious medical condition, laboratory abnormalities, or psychiatric disorder, that in the opinion of the Investigator places the patients at unacceptable risk if he/she were to participate in the study.
* Clinically relevant active infection including active hepatitis B or C, Human Immunodeficiency Virus (HIV) infection, or any other concurrent disease which, in the judgment of the Investigator, would make the patients inappropriate for enrollment into this study.
* Significant cardiac disease such as recent myocardial infarction (≤ 6 months prior to Day 1), unstable angina, uncontrolled congestive heart failure, uncontrolled hypertension (recurrent or persistent increases in systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg ), uncontrolled cardiac arrhythmias, grade 3 or greater cardiac toxicity following prior chemotherapy.
* History of multiple sclerosis or other demyelinating disease, Eaton-Lambert syndrome (para-neoplastic syndrome), history of hemorrhagic or ischemic stroke within the last 6 months, central nervous system (CNS) injury with residual neurological deficit, or alcoholic liver disease.
* Treatment with another investigational agent during the study or ≤ 4 weeks prior to Day 1.
* Prior malignancy within the last 3 years except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer.
* Patients who have any known recent biochemical or clinical evidence of pancreatitis or extensive metastatic disease involving the pancreas that is associated with an increased amylase and/or lipase will be excluded. (Note: Enrollment of patients with any metastatic disease to, or around, the pancreas may be allowed only with agreement between the Sponsor and the Investigator).
* WCBP who are pregnant or breast feeding or men and women not using adequate contraception are excluded.
* Patients unwilling or unable to comply with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-12; Primary Completion 2013-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Determine the MTD/RPTD and response rate To assess the response rate of the combination at the MTD, in the patient population | during study

SECONDARY OUTCOMES:
Objective response rate (OR and CR), duration of responses, time to progression, progression-free survival, and overall survival and pharmacodynamics. | during the study

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Southern California, Los Angeles, California
  - Comprehensive Cancer Center of the Desert, Palm Springs, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - CTRC at University of Texas Health Science Center, San Antonio, Texas